CLINICAL TRIAL: NCT03673683
Title: Sedation AND Weaning in Children: the SANDWICH Trial
Brief Title: Sedation and Weaning in Children Requiring Invasive Mechanical Ventilation
Acronym: SANDWICH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Collaborators: Birmingham Women's and Children's NHS Foundation Trust (Other); Royal Brompton & Harefield NHS Foundation Trust (Other); University College, London (Other); University of Birmingham (Other); University of Leeds (Other); Northern Ireland Clinical Trials Unit (Other); University of the West of England (Other); University of Edinburgh (Other)
Responsible Party: Principal Investigator, Bronagh Blackwood, Professor, Queen's University, Belfast
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: B17/13; 15/04/01 (Other: NIHR HTA)
Record Dates: First submitted 2018-07-02; First posted 2018-09-17 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Ventilator Weaning
Keywords: Invasive Mechanical Ventilation

STUDY DESIGN:
Intervention Model Description: Stepped wedge, cluster randomized stepped wedge clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator): Sedation and ventilation weaning that is non-protocol-based and primarily medically-driven.
  Interventions: Behavioral: Usual care
- SANDWICH protocol (Experimental): A protocol-based intervention for managing sedation and ventilation weaning.
  Interventions: Behavioral: SANDWICH protocol

INTERVENTIONS:
Behavioral: SANDWICH protocol — A protocol based intervention incorporating co-ordinated care with greater nursing involvement; patient-relevant sedation plans linked to regular assessment using the COMFORT scale; regular assessment of ventilation parameters with a higher than usual trigger for undertaking an extubation readiness test; a spontaneous breathing trial (SBT) on low levels of respiratory support to test extubation readiness
  Arms: SANDWICH protocol
Behavioral: Usual care — Usual sedation and weaning management that is not protocol based
  Arms: Usual Care

SUMMARY:
A UK multi-centre cluster randomised controlled trial to determine if a protocol-based intervention incorporating coordinated care with greater nursing involvement to managing sedation and ventilator weaning can reduce the duration of invasive mechanical ventilation and is cost effective compared with usual care in children in Pediatric Intensive Care Units.

DETAILED DESCRIPTION:
Mechanical ventilation is a common lifesaving therapy, but the longer a child remains on the ventilator, the more risk they have of developing problems. For this reason, getting the child off the ventilator (called weaning) is an important patient outcome. Sedative drugs are necessary so the child can tolerate the breathing tube, but too much can make them sleepy and delay coming off the ventilator.

In 2014, visits to 24 Paediatric Intensive Care Units (PICUs) were conducted and it was found that weaning was usually performed by doctors and occasionally senior nurses, but weaning was not always done the same way and, because everyone was not involved, it was often disjointed.

This study will determine if a coordinated approach by doctors and nurses to optimise sedation and weaning using guidelines will: (a) reduce how long patients are on a ventilator without causing any increased risk; (b) reduce the time children spend in a PICU and the hospital; (c) be cost effective in the NHS; and (d) be easily adopted by staff delivering care.

Children receiving ventilation, except those that will never come off a ventilator, will be weaned using the guidelines. Data collection will start in all PICUs at the same time from the very beginning of the study when they are weaning children according to usual practice. Each month, one unit will be chosen at random and staff will be trained to use the new guidelines. The unit will continue using the new guidelines for the rest of the trial. Outcome data collected before (usual care) and after (intervention) training will be compared. An evaluation of the process of implementing the new intervention will be undertaken. During the process evaluation, study staff will be interviewed about their experiences and views with the new approach.

ELIGIBILITY:
Inclusion Criteria:

* All children (> 16 year old) in participating PICUs receiving invasive mechanical ventilation

Exclusion Criteria:

* Children who would not reach the primary endpoint (tracheostomy in situ; not expected to survive; treatment withdrawal)
* Children who are pregnant, as documented in their medical notes

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10498 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Duration of Invasive Mechanical Ventilation | From admission until 48 hours following extubation
  Duration of Invasive Mechanical Ventilation measured in hours from initiation of invasive mechanical ventilation until the first successful extubation

SECONDARY OUTCOMES:
Successful Extubation | 48 hours following extubation
  Incidence of successful extubation
Number of unplanned extubations | From admission up to 90 days or PICU discharge whichever is earlier
  Number of unplanned extubations
Number of reintubations | From admission up to 90 days or PICU discharge whichever is earlier
  Number of reintubations
Total duration of Invasive mechanical ventilation | From admission up to 90 days or PICU discharge whichever is earlier
  Total duration of Invasive mechanical ventilation
Non-invasive mechanical ventilation Incidence | From admission up to 90 days or PICU discharge whichever is earlier
  Incidence of post-extubation use of non-invasive ventilation
Non-invasive mechanical ventilation Duration | From admission up to 90 days or PICU discharge whichever is earlier
  Duration of post-extubation use of non-invasive ventilation
Tracheostomy insertion | From admission up to 90 days or PICU discharge whichever is earlier
  Incidence of tracheostomy insertion
Post-extubation stridor | From admission up to 90 days or PICU discharge whichever is earlier
  Incidence of post-extubation stridor
Adverse events | From admission up to 90 days or PICU discharge whichever is earlier
  Incidence of adverse events
PICU length of stay | From admission up to 90 days or PICU discharge whichever is earlier
  PICU length of stay from admission to discharge measured in days
Hospital length of stay | From admission up to 90 days or PICU discharge whichever is earlier
  Hospital length of stay from admission to discharge measured in days
ICU Mortality | From admission up to 90 days or PICU discharge whichever is earlier
  Incidence of mortality occurring within the ICU
Hospital Mortality | From admission up to 90 days or PICU discharge whichever is earlier
  Incidence of Mortality occurring within the hospital
Cost per respiratory complication avoided | 28 days
  Cost per respiratory complication avoided

CONTACTS AND LOCATIONS:
Overall Officials: Bronagh Blackwood, Principal Investigator — Queens University Belfast
Locations (17):
- United Kingdom (17):
  - Belfast Health and Social Care Trust, Belfast, Co. Antrim
  - Alder Hey Children's NHS Foundation Trust, Liverpool, Merseyside
  - University Hospitals of North Midlands NHS Trust, Stoke, Staffordshire
  - Birmingham Women and Children's NHS Foundation Trust, Birmingham
  - University Hospital Bristol NHS Foundation Trust, Bristol
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Cardiff and Vale University Health Board, Cardiff
  - Leeds Teaching Hospitals Trust, Leeds
  - Kings College Hospital NHS Foundation Trust, London
  - St George's University Hospitals NHS Foundation Trust, London
  - Royal Brompton and Harefield NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London
  - Great Ormond Street Hospital NHS Foundation Trust, London
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle
  - Oxford University Hospital NHS Foundation Trust, Oxford
  - Sheffield Children's NHS Foundation Trust, Sheffield
  - University Hospital Southampton Foundation NHS Trust, Southampton